CLINICAL TRIAL: NCT00386763
Title: A Randomized, Investigator-Blinded, Multicenter, Parallel-Group Study to Compare Efficacy, Safety and Tolerability of Arthemeter/ Lumefantrine Dispersible Tablet Formulation vs. Artemether/ Lumefantrine 6-Dose Crushed Tablet in the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in Infants and Children.
Brief Title: Efficacy and Safety of the Pediatric Formulation of Artemether- Lumefantrine in Children With Uncomplicated P. Falciparum Malaria.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCOA566B2303
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Malaria; Falciparum
Keywords: Marsh fever; Plasmodium infections; Remittent fever; Paludism; Artemether; Artemisinins; Malaria; Benflumetol; Lumefantrine
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: Artemether-lumefantrine

SUMMARY:
This study will evaluate the safety and efficacy of artemether-lumefantrine against uncomplicated malaria caused P. falciparum in children of 5-35 kg bodyweight.

ELIGIBILITY:
Inclusion Criteria:

* male or female infants and children ≤12 years of age
* body weight of ≥5 kg and <35 kg,
* with a confirmed diagnosis of uncomplicated malaria caused by the P. falciparum parasite

Exclusion Criteria:

* complicated malaria
* persistent vomiting
* malaria due to parasites other than P. falciparum
* antimalarial treatment received in the past 2 weeks
* known chronic disease e.g. positive HIV status, severe cardiac, renal, or hepatic disease

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 890
Dates: Start 2006-08; Study Completion 2007-03

PRIMARY OUTCOMES:
Proportion of patients free of parasites at day 28.

SECONDARY OUTCOMES:
Proportion of patients free of parasites at 7 days and at 14 days
Time to clearance from parasites
Time to clearance of fever
Hematology and biochemistry parameters
Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (5):
- Novartis, Benin, Benin
- Novartis, Kenya, Kenya
- Novartis, Mali, Mali
- Novartis, Mozambique, Mozambique
- Novartis, Tanzania, Tanzania

REFERENCES:
- [Derived] Belard S, Ramharter M, Kurth F. Paediatric formulations of artemisinin-based combination therapies for treating uncomplicated malaria in children. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD009568. doi: 10.1002/14651858.CD009568.pub2. PMID 33289099
- [Derived] Abdulla S, Sagara I, Borrmann S, D'Alessandro U, Gonzalez R, Hamel M, Ogutu B, Martensson A, Lyimo J, Maiga H, Sasi P, Nahum A, Bassat Q, Juma E, Otieno L, Bjorkman A, Beck HP, Andriano K, Cousin M, Lefevre G, Ubben D, Premji Z. Efficacy and safety of artemether-lumefantrine dispersible tablets compared with crushed commercial tablets in African infants and children with uncomplicated malaria: a randomised, single-blind, multicentre trial. Lancet. 2008 Nov 22;372(9652):1819-27. doi: 10.1016/S0140-6736(08)61492-0. Epub 2008 Oct 14. PMID 18926569